CLINICAL TRIAL: NCT04266522
Title: Medical Physics Direct Patient Care Initiative - Communication Intervention Study Protocol
Brief Title: Medical Physics Direct Patient Care for the Improvement of Patient Understanding of Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jay Burmeister, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-104; P30CA022453 (NIH)
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (printed materials) (Active Comparator): Patients receive printed materials describing the technical aspects of their treatment.
  Interventions: Other: Informational Intervention; Other: Questionnaire Administration
- Arm II (printed materials, physicist interaction) (Experimental): Patients receive printed materials as in Arm I. Patients also receive a minimum of 2 direct physicist interactions to describe the technical aspects of their treatment either immediately prior to or immediately after treatment simulation.
  Interventions: Other: Informational Intervention; Other: Counseling; Other: Questionnaire Administration

INTERVENTIONS:
Other: Informational Intervention — Receive printed materials
Other: Counseling — Receive direct physicist interactions to describe the technical aspects of the treatment
  Other Names: counseling, Counseling Intervention
  Arms: Arm II (printed materials, physicist interaction)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well medical physics direct patient care works in improving patients' understanding of their cancer treatment. Providing direct physicist-patient interactions and answering patients' questions about their cancer treatment may help patients to understand the care and therefore reduce anxiety and distress during treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate whether the Medical Physics Direct Patient Care Initiative (MPDPCI) improves anxiety/distress.

SECONDARY OBJECTIVE:

II. To assess whether the MPDPCI improves patient treatment adherence and overall satisfaction.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive printed materials describing the technical aspects of their treatment.

ARM II: Patients receive printed materials as in Arm I. Patients also receive a minimum of 2 direct physicist interactions to describe the technical aspects of their treatment either immediately prior to or immediately after treatment simulation.

ELIGIBILITY:
Inclusion Criteria:

* Medical physicists will be eligible if they care for patients within the Gershenson Radiation Oncology Center within the Karmanos Cancer Institute and have completed the patient communication training
* Are able to read and write in English
* Are scheduled for curative radiation therapy at the Gershenson Radiation Oncology Center

Exclusion Criteria:

* NONE

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Anxiety | 4 months
  Will be assessed using linear mixed-effects models. These objectives will be evaluated based on the difference between groups across three time points (i.e., group-effect) using the baseline corrected measurements. Each patient will be considered as random-effects along with the repeated measurements at three time points. The repeated measurements at three time points will be handled by autocorrelated residuals within groups.
Distress | 4 months
  Will be assessed using linear mixed-effects models. These objectives will be evaluated based on the difference between groups across three time points (i.e., group-effect) using the baseline corrected measurements. Each patient will be considered as random-effects along with the repeated measurements at three time points. The repeated measurements at three time points will be handled by autocorrelated residuals within groups.

SECONDARY OUTCOMES:
Patient treatment adherence | 4 months
  Will be assessed using 2-sided unpaired t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Burmeister, PhD, Principal Investigator — Barbara Ann Karmanos Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No